CLINICAL TRIAL: NCT00513370
Title: A Canadian Open-Label Access Program to Evaluate the Safety and the Effectiveness of Adalimumab When Added to Inadequate Therapy for the Treatment of Psoriasis
Brief Title: A Canadian Open-Label Access Program to Evaluate Adalimumab When Added to Inadequate Therapy for the Treatment of Psoriasis
Acronym: PRIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Isabel Pereira, Affiliate Project Manager, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W10-151
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; adalimumab
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Humira (adalimumab)

INTERVENTIONS:
Biological: Humira (adalimumab) — Study drug will be provided as a sterile, preservative-free solution for subcutaneous injection, contained in a pre-filled syringe housed in a pen device (pre-filled pen). Loading dose of 80 mg of adalimumab subcutaneously (sc) at Baseline, and 40 mg of adalimumab sc at Week 1, followed by 40 mg of adalimumab sc every other week (eow) for 24 weeks.
  Other Names: ABT-D2E7; adalimumab; Humira

SUMMARY:
To evaluate the safety profile, the effectiveness and the economic impact of adalimumab when used for the treatment of subjects with active plaque psoriasis who have not adequately responded to prior psoriasis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of psoriasis for at least 6 months prior to the Screening, as determined by subject interview of his/her medical history and confirmation of diagnosis through physical examination by the investigator
* Subject must have stable plaque psoriasis for at least 2 months prior to the Screening, as determined by subject interview of his/her medical history
* Subject has moderate to severely active plaque psoriasis at Baseline defined as: BSA (Body Surface Area) > 10% and a Psoriasis Area and Severity Index (PASI) > 12
* Subject has active psoriasis despite treatment with topical agents
* Subject has failed to respond to, is intolerant to or unable to access phototherapy
* Subject has failed to respond to, is intolerant to or has contraindication for at least two of the following therapies:

  * CyA (Cyclosporine A)
  * MTX (Methotrexate)
  * Oral retinoid
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:

  * Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)
  * Contraceptives (oral or parenteral) for three months (90 days) prior to study drug administration
  * A vasectomized partner
  * Total abstinence from sexual intercourse
* If female and of childbearing potential, the result of a serum pregnancy test performed at Screening is negative
* Able and willing to self-administer sc injections or has available qualified person(s) to administer sc injections
* Able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

* Subject has other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with the evaluation of psoriasis or compromise the subject's safety
* Subject has erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis as the primary morphology of their psoriasis
* Subject has a history of an allergic reaction or significant sensitivity to constituents of adalimumab
* Investigational agents not mentioned must be discontinued at least 30 days or 5 half-lives prior to the Baseline visit (whichever is longer)
* Topical therapies:

  * Subject started receiving a new topical therapy within the last four weeks prior to the Baseline visit for areas other than the palms, soles of feet, axilla and groin.
  * Dose(s) and regimen(s) of topical therapy(ies) that the subject is receiving at the Baseline visit, for areas other than the palms, soles of feet, axilla and groin, was (were) increased during the four weeks that preceded the Baseline visit.
  * Subject is likely to require the initiation of a new topical therapy for the treatment of psoriasis such as corticosteroids, vitamin D analogs, or retinoids during the first 16 weeks that will follow the Baseline visit. (During the first 16 weeks that will follow the Baseline visit, initiation of topical therapies are allowed for the palms, soles of feet, axilla and groin area only).
* Oral or injectable corticosteroids therapies:

  * Subject started receiving oral or injectable doses of corticosteroids within the last four weeks prior to the Baseline visit.
  * Dose(s) and regimen(s) of corticosteroids therapy(ies) that the subject is receiving at the Baseline visit, was (were) increased during the four weeks that preceded the Baseline visit.
  * Subject is likely to require the initiation of oral or injectable dose of corticosteroids therapies for the treatment of psoriasis during the first 16 weeks that will follow the Baseline visit.
* Phototherapies

  * Subject started being treated with UVB phototherapy, within the last four weeks prior to the Baseline visit.
  * Regimen(s) of concomitant UVB phototherapy that the subject is receiving at the Baseline visit was (were) increased during the four weeks that preceded the Baseline visit.
  * Subject is likely to require the initiation of UVB therapy during the first 16 weeks that will follow the Baseline visit.
  * Subject was treated with psoralen UVA (PUVA) phototherapy within the last four weeks prior to the Baseline visit.
  * Subject is likely to require PUVA phototherapy during the course of the study.
  * Subject cannot avoid excessive sun exposure or the use of tanning booths for at least 2 weeks prior to Baseline and during the first 16 weeks that will follow the Baseline visit.
* Systemic Therapies:

  * Subject has been initiated on a new systemic agent for the treatment of psoriasis within the last four weeks prior to the Baseline visit.
  * Dose(s) and regimen(s) of systemic therapy(ies) that the subject is receiving at the Baseline visit, was (were) increased during the four weeks that preceded the Baseline visit.
  * Subject is likely to require the initiation of systemic therapy, other than adalimumab, for the treatment of psoriasis during the first 16 weeks that will follow the Baseline visit.
  * Subject has been treated with systemic calcineurin inhibitors (cyclosporin, FK506 and others) within the last four weeks prior to the Baseline visit.
  * Subject is likely to receive systemic calcineurin inhibitors during the course of the study.
  * Subject has received Anakinra/Kineret within the last 2 weeks prior to the Baseline visit and is likely to receive Anakinra/Kineret during the course of the study.
* Subject cannot discontinue the following systemic psoriasis therapies:

  * Alefacept must be discontinued at least 12 weeks prior to the Baseline visit.
  * Efalizumab must be discontinued at least 6 weeks prior to the Baseline visit.
  * Infliximab must be discontinued at least 8 weeks prior to the Baseline visit.
  * Etanercept must be discontinued at least 3 weeks prior to the Baseline visit.
* Subject has a history of cancer or lymphoproliferative disease other than:

  * Successfully and completely treated Cervical dysplasia, with no recurrence within the last five years.
* Has a history of uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure, New York Heart Association (NYHA) III, IV, recent stroke (within three months), chronic leg ulcer and any other condition (e.g., indwelling urinary catheter) which, in the opinion of the Investigator, would put the subject at risk by participation in the protocol or who would make the subject unsuitable for the study.
* Positive serology for hepatitis B indicating acute or chronic infection.
* Currently taking or likely to begin anti-retroviral therapy at any time during the course of the study.
* Subject is known to have immune deficiency, history of human immunodeficiency virus (HIV) or is immunocompromised.
* Persistent or recurrent or severe infections requiring hospitalization or treatment with intra-venous (IV) antibiotics within 30 days, or oral antibiotics within 14 days, prior to Baseline.
* Female subjects who are pregnant or breastfeeding.
* Has a history of clinically significant drug or alcohol abuse in the last year.
* Previous diagnosis or signs of central nervous system demyelinating diseases (e.g., optic neuritis, visual disturbance, gait disorder/ataxia, facial paresis, apraxia).
* History of active tuberculosis (TB), history of histoplasmosis or listeriosis.
* Has latent TB (positive purified protein derivative (PPD) skin test, two-step PPD when applicable, and chest X-ray indicative of TB) or has other risk factors for the activation of latent TB, e.g. previous exposure to TB, and has not initiated TB prophylaxis prior to the first adalimumab treatment. In either case, the Abbott Medical Advisor must be contacted before initiating the study treatment.
* Subjects will be excluded if the CXR is found to have changes suggestive of old healed tuberculous lesion (e.g. calcified nodule, fibrotic scar, apical or basilar pleural thickening etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Papp, MD PhD FRCPC, Principal Investigator — K. Papp Clinical Research Inc.
Locations (22):
- Canada (22):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Fenwick, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Markham, Ontario
  - Nepean, Ontario
  - North Bay, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
  - Ste-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab 40 mg Eow: adalimumab 40 mg every other week (eow)
Period: Overall Study
Arm/Group | Adalimumab 40 mg Eow
Started | 203
Completed | 179
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 192
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 124
Region of Enrollment [Number; unit: participants]
  Canada | 203

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Psoriasis Area and Severity Index (PASI) 75 Response at 16 Weeks
Description: PASI 75 is a 75% or greater improvement on the Psoriasis Area and Severity Index (PASI). The PASI scale runs from 0-72, where 0 = no psoriasis and 72 = complete erythroderma of the severest possible degree
Time Frame: 16 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Number; unit: participants
Groups:
- Adalimumab 40 mg Eow - 16 Weeks: adalimumab 40 mg every other week - Week 16 timepoint
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks
Number analyzed (Participants) | 191
participants
  Responder | 144
  Non-responder | 47

2. Secondary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at 16 and 24 Weeks
Description: Mean change in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI score ranges from 0-72, where 0 = no psoriasis and 72 = complete erythroderma of the severest possible degree
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: unit on a scale
Groups:
- Adalimumab 40 mg Eow - 24 Weeks: adalimumab 40 mg every other week - Week 24 timepoint
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 191 | 183
unit on a scale
  Change from Baseline | -15.9 (7.55) | -16.1 (7.46)

3. Secondary Outcome: Mean Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at 16 and 24 Weeks
Description: Mean percent change in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI score ranges from 0-72, where 0 = no psoriasis and 72 = complete erythroderma of the severest possible degree.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Adalimumab 40 mg Eow - 24 Weeks: adalimumab 40 mg every other week - Week 16 timepoint
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 191 | 183
percent change | -81.5 (23.63) | -83.0 (23.47)

4. Secondary Outcome: Number of Subjects With Improvement in Physician's Global Assessment for Psoriasis (PGA)
Description: Number of subjects with improvement on the Physician's Global Assessment for Psoriasis (PGA). The PGA is a 6-point scale used to measure the severity of disease at the time of the physician's evaluation of the subject, where 0 = clear and 6 = very severe. Improvement is defined as a reduction in PGA score.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 203 | 181
participants | 174 | 164

5. Secondary Outcome: Number of Subjects Achieving a Clinical Response Defined as a Physician's Global Assessment for Psoriasis (PGA) of "Clear" or "Clear or Minimal"
Description: Number of subjects achieving a response of "Clear" or "Clear or Minimal" on the Physician's Global Assessment for Psoriasis. This is a 6-point scale used to measure the severity of disease at the time of the physician's evaluation of the subject. The degree of overall severity is rated as follows: 0-Clear, 1-Minimal, 2-Mild, 3-Moderate, 4-severe, 5-very severe.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 191 | 183
participants
  Subjects achieving "Clear" | 53 | 59
  Subjects achieving "Clear or Minimal" | 111 | 121

6. Secondary Outcome: Mean Change From Baseline in Physician Global Assessment of Arthritic Disease Activity at 16 and 24 Weeks
Description: Mean Change from Baseline in Physician Global Assessment of Arthritic Disease Activity as measured on a 100-mm visual analog scale where 0 mm = no arthritis activity and 100 mm = extremely active arthritis.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 91 | 85
units on a scale | -18.7 (23.48) | -20.9 (23.32)

7. Secondary Outcome: Number of Subjects With Psoriasis Area and Severity Index (PASI) 50/75/90/100 Response
Description: PASI 50/75/90/100 is a >=50% / >=75% / >=90% / 100% improvement on the Psoriasis Area and Severity Index (PASI). The PASI scale runs from 0-72, where 0 = no psoriasis and 72 = complete erythroderma of the severest possible degree.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 191 | 183
participants
  Subjects achieving PASI 50 | 169 | 163
  Subjects achieving PASI 75 | 144 | 140
  Subjects achieving PASI 90 | 100 | 102
  Subjects achieving PASI 100 | 49 | 58

8. Secondary Outcome: Mean Change From Baseline in Tender Joint Count at 16 and 24 Weeks
Description: Mean change in the number of tender joints from Baseline. 78 joints were evaluated for tenderness, including all 76 joints evaluated for swelling plus the hip joints.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: number of joints
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 40 | 39
number of joints | -8.7 (13.57) | -8.7 (14.83)

9. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count at 16 and 24 Weeks
Description: Mean change in the number of swollen joints from Baseline. 76 joints were evaluated for swelling, corresponding to all joints evaluated for tenderness except for the hip joints.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: number of joints
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 31 | 31
number of joints | -4.7 (5.35) | -4.9 (7.08)

10. Secondary Outcome: Mean Change From Baseline in Patient's Global Assessment of Joint Pain at 16 and 24 Weeks
Description: Mean change in the Patient's Global Assessment of Joint Pain from Baseline, as assessed on a 100-mm visual analog scale where 0 mm = no pain and 100 mm = pain as bad as it could be.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 137 | 129
units on a scale | -20.9 (31.77) | -19.3 (32.02)

11. Secondary Outcome: Mean Change From Baseline in the Dermatology Life Quality Index (DLQI) at 16 and 24 Weeks
Description: Mean change in the Dermatology Life Quality Index (DLQI) from Baseline. The questionnaire contains 10 questions and is scored from 0-30, where 0 = total lack of impairment and 30 = my life is very much impaired; the minimum clinically important difference is 2.3 to 5.7 point change.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 191 | 182
units on a scale | -9.8 (7.09) | -10.1 (7.26)

12. Secondary Outcome: Number of Subjects Achieving a Dermatology Life Quality Index (DLQI) = 0
Description: Number of subjects achieving a Dermatology Life Quality Index (DLQI) score of 0 (indicating total lack of impairment). The DLQI consists of 10 questions and is scored from 0-30, where 0 = total lack of impairment and 30 = my life is very much impaired.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 191 | 182
participants | 67 | 83

13. Secondary Outcome: Mean Change From Baseline in Beck Depression Inventory (BDI-II) at 16 and 24 Weeks
Description: Change in the Beck Depression Inventory from Baseline. The BDI-II contains 21 questions and is scored from 0-63; higher scores indicate more severe depression symptoms.
Time Frame: 16 and 24 weeks
Population: Observed Cases - subjects with nonmissing values at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg Eow - 16 Weeks | Adalimumab 40 mg Eow - 24 Weeks
Number analyzed (Participants) | 175 | 173
units on a scale | -4.1 (6.56) | -4.3 (6.71)

14. Secondary Outcome: Change From Baseline on the EuroQol (EQ-5D) Quality of Life Questionnaire
Time Frame: 16 and 24 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: units on a scale

15. Secondary Outcome: Change in Productivity Outcomes and Costs From Baseline as Measured by the Health and Labour Questionnaire (HLQ)
Time Frame: 16 and 24 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: units on a scale

16. Secondary Outcome: Change in Resource Utilization Outcomes and Costs From Baseline as Measured by the Health Care Resource (HCR) Questionnaire
Time Frame: 16 and 24 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: units on a scale

ADVERSE EVENTS:
Arm/Group | Adalimumab 40 mg Eow
Serious Adverse Events (participants affected / at risk) | 9
Other Adverse Events (participants affected / at risk) | 145
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Adalimumab 40 mg Eow
Tongue oedema (Gastrointestinal disorders) | 1/203 (1)
Myocardial infarction (Cardiac disorders) | 2/203 (2)
Pericarditis (Cardiac disorders) | 1/203 (1)
Death (General disorders) | 1/203 (1)
Appendicitis (Infections and infestations) | 1/203 (1)
Pneumonia (Infections and infestations) | 1/203 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/203 (1)
Renal vasculitis (Renal and urinary disorders) | 1/203 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1/203 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Adalimumab 40 mg Eow
Diarrhoea (Gastrointestinal disorders) | 6/203 (7)
Nausea (Gastrointestinal disorders) | 6/203 (6)
Injection site reaction (General disorders) | 7/203 (10)
Fatigue (General disorders) | 5/203 (5)
Oedema peripheral (General disorders) | 5/203 (5)
Injection site erythema (General disorders) | 4/203 (16)
Upper respiratory tract infection (Infections and infestations) | 22/203 (30)
Nasopharyngitis (Infections and infestations) | 22/203 (24)
Influenza (Infections and infestations) | 10/203 (12)
Bronchitis (Infections and infestations) | 6/203 (6)
Pharyngitis (Infections and infestations) | 5/203 (5)
Gastroenteritis (Infections and infestations) | 5/203 (5)
Pneumonia (Infections and infestations) | 4/203 (4)
Sinusitis (Infections and infestations) | 4/203 (5)
Pharyngitis streptococcal (Infections and infestations) | 4/203 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8/203 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 5/203 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/203 (5)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 4/203 (4)
Headache (Nervous system disorders) | 10/203 (16)
Migraine (Nervous system disorders) | 4/203 (4)
Dizziness (Nervous system disorders) | 4/203 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5/203 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4/203 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 7/203 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 6/203 (7)
Hypertension (Vascular disorders) | 7/203 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication and presentation of this Study shall reside with Abbott. No independent manuscript may be submitted for publication until the first manuscript has been accepted for publication or twelve (12) months after completion of Study at all sites, which ever occurs first.